CLINICAL TRIAL: NCT00218816
Title: Nebulizer Intervention for Minority Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Arlene Butz, ScD, RN, MSN, Professor, Johns Hopkins University School of Medicine Department of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 99-01-06-02; 5R01NR005060-04 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-09-05 (Estimated); Status verified 2008-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Nebulizer Education Intervention
- 2 (Other)
  Interventions: Behavioral: Standard Asthma Education Groups

INTERVENTIONS:
Behavioral: Nebulizer Education Intervention — Asthma Education
  Arms: 1
Behavioral: Standard Asthma Education Groups — Asthma Education
  Arms: 2

SUMMARY:
To determine if teaching parents and children to identify the child's asthma symptoms early and if teaching the appropriate use of a nebulizer will result in a decrease in emergency department visits.

DETAILED DESCRIPTION:
Nebulizer use in young children is common with prevalence of 33-71% in children under age 12 years. Nebulizers are used primarily to administer SABA medications, (i.e., albuterol) and some anti-inflammatory medications (i.e., budesonide, cromolyn). Parents may prefer nebulizer delivery due to the inability of young children to coordinate respiration with aerosol delivery and many parents lack confidence in administering metered-dose inhaler (MDI) medications to young children. Physician preference for nebulizer administration of asthma medications is low, but is favored due to direct medication delivery to the respiratory system despite studies indicating MDIs with spacers are as effective as nebulizers in delivering asthma medications to young children. Although national guidelines recommend a nebulizer with mask for children 2 years or younger most asthma educational programs lack specific content addressing appropriate nebulizer technique including when and what symptoms to treat at home, optimal length of a nebulized medication session, prevention of SABA overuse and appropriate cleaning and maintenance of the device. Because the overuse of home nebulizer SABA medications has been associated with fatal asthma, instruction and supervision of nebulized rescue medication delivery in addition to appropriate preventive medication use may reduce asthma morbidity and mortality .

The current study was conducted to determine the effectiveness of a home-based nebulizer educational intervention (NEI) for young children with asthma. The intervention was designed to teach early symptom recognition, appropriate medication use and nebulizer technique for home treatment of acute asthma episodes. Study outcomes included symptom frequency, activity limitation, emergency department (ED) visits and hospitalizations, appropriate asthma medication use and nebulizer practice. We hypothesized that children receiving the NEI would demonstrate improvement in appropriate nebulizer and asthma medication use and decreased asthma symptoms, activity limitation, ED visits and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed asthma, use of nebulizer in past 30 days, wheezing or cough symptoms at least weekly during the past 30 days.

Exclusion Criteria:

* Participation in another asthma study or having other respiratory illness such as cystic fibrosis, BPD

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2000-08; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
We hypothesized that children receiving the NEI would demonstrate improvement in appropriate nebulizer and asthma medication use and decreased asthma symptoms, activity limitation, ED visits, and hospitalizations. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Arlene M Butz, SCD,MSN,BSN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Butz AM, Huss K, Mudd K, Donithan M, Rand C, Bollinger ME. Asthma management practices at home in young inner-city children. J Asthma. 2004 Jun;41(4):433-44. doi: 10.1081/jas-120033985. PMID 15281329
- [Background] Butz AM, Donithan M, Bollinger ME, Rand C, Thompson RE. Monitoring nebulizer use in children: comparison of electronic and asthma diary data. Ann Allergy Asthma Immunol. 2005 Mar;94(3):360-5. doi: 10.1016/S1081-1206(10)60988-X. PMID 15801247
- [Background] Butz AM, Syron L, Johnson B, Spaulding J, Walker M, Bollinger ME. Home-based asthma self-management education for inner city children. Public Health Nurs. 2005 May-Jun;22(3):189-99. doi: 10.1111/j.0737-1209.2005.220302.x. PMID 15982192